CLINICAL TRIAL: NCT03020238
Title: Impact of Nerve-sparing Radical Hysterectomy on Patients' Urinary Dynamics: a Randomized Controlled Trial
Brief Title: Impact of Nerve-sparing Radical Hysterectomy on Patients' Urinary Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, Associate Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-OBGYN-2013
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Cancer; Urinary Retention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BiClamp group (Placebo Comparator): BiClamp forcep (BiClamp® forcep, ERBE Elektromedizin, GmbH, Tuebingen, Germany) is used to dissect inferior hypogastric plexus
  Interventions: Procedure: BiClamp group
- water jet group (Active Comparator): water jet (ERBEJET®2, ERBE Elektromedizin, GmbH, Tuebingen, Germany) is used to dissect inferior hypogastric plexus
  Interventions: Procedure: water jet group

INTERVENTIONS:
Procedure: BiClamp group — electric energy
  Other Names: BiClamp® forcep, ERBE Elektromedizin
  Arms: BiClamp group
Procedure: water jet group — water jet energy
  Other Names: ERBEJET®2, ERBE Elektromedizin
  Arms: water jet group

SUMMARY:
Background: Radical hysterectomy is an important therapy for early cervical cancer. Disfunction of urinary dynamics is the most common postoperative adverse effects, which had negative impact on patients' quality of life. Nerve sparing radical hysterectomy (NSRH) could reserve inferior hypogastric plexus (IHP) innervating bladder, hence improving postoperative urinary dynamics. Furthermore impact of different energy instruments on urinary dynamic isn't clear.

Objectives: This study is to compare urinary dynamics before and after NSRH, and to analyze the difference between BiClamp forcep (BiClamp® forcep, ERBE Elektromedizin, GmbH, Tuebingen, Germany) and water jet (ERBEJET®2) about the effects of dissecting IHP.

Study population: Cervical cancer of FIGO IB stage, among which 120 cases are enrolled to randomly allocated to BiClamp group or water jet group.

Intervention: Patients accept NSRH which all will be accomplished by Professor Ming Wu.

Methods: All surgical patients are accessed via urinary dynamics before and four months after NSRH. On the 14th day after surgeries, urinary catheter will be removed and residual urine volume (RUV) will be measured. For patients of RUV > 100 ml, urinary catheter will be replaced.

Primary study endpoint: the successful rate of removing urinary catheter on the 14th day after NSRH.

Secondary study endpoint: urinary dynamics four months after NSRH.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage IB
* ASA score 0-2

Exclusion Criteria:

* Radiotherapy or chemotherapy before surgeries
* ASA score > 2
* With abnormal urinary dynamics before surgeries

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
successful rate of removing urinary catheter | 14th day after nerve-sparing radical hysterectomy
  successful rate (%) of removing urinary catheter assessed by residual urine volume less than 100 ml

SECONDARY OUTCOMES:
urinary dynamics parameters determined by urodynamics apparatus: bladder capacity and sensation | four months after nerve-sparing radical hysterectomy
  bladder capacity and sensation in ml
urinary dynamics parameters determined by urodynamics apparatus: residual urine volume | four months after nerve-sparing radical hysterectomy
  residual urine volume in ml
urinary dynamics parameters determined by urodynamics apparatus: urine flow rate | four months after nerve-sparing radical hysterectomy
  urine flow rate in ml/s
urinary dynamics parameters determined by urodynamics apparatus: bladder pressure | four months after nerve-sparing radical hysterectomy
  bladder pressure in cmH2O
urinary dynamics parameters determined by urodynamics apparatus: detrusor pressure | four months after nerve-sparing radical hysterectomy
  detrusor pressure in cmH2O
urinary dynamics parameters determined by urodynamics apparatus: bladder compliance | four months after nerve-sparing radical hysterectomy
  bladder compliance in ml/cmH2O
survival outcomes: ovarall survival | two years after nerve-sparing radical hysterectomy
  overall survival in months
survival outcomes: progression-free survival | two years after nerve-sparing radical hysterectomy
  progression-free survival in months

CONTACTS AND LOCATIONS:
Overall Officials: Wu Ming, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with authorised researchers via online database.